CLINICAL TRIAL: NCT01522443
Title: A Phase 3, Randomized, Double-blind, Controlled Trial of Cabozantinib (XL184) Versus Mitoxantrone Plus Prednisone in Men With Previously Treated Symptomatic Castration-resistant Prostate Cancer
Brief Title: Study of Cabozantinib (XL184) Versus Mitoxantrone Plus Prednisone in Men With Previously Treated Symptomatic Castration-resistant Prostate Cancer
Acronym: COMET-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped after the outcome of cabozantinib Phase 3 CRPC study XL184-307.
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL184-306
Record Dates: First submitted 2012-01-13; First posted 2012-01-31 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer; Castration Resistant Prostate Cancer; Pain; Prostatic Neoplasms
Keywords: prostate cancer; castration resistant prostate cancer; bone pain; CRPC
MeSH Terms: conditions — Prostatic Neoplasms; Pain | interventions — cabozantinib; Mitoxantrone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabozantinib (Experimental): Subjects randomized to the cabozantinib arm will also receive placebo mitoxantrone injections (color-matched with methylene blue) and placebo prednisone capsules.
  There will be a maximum of 10 infusions for mitoxantrone placebo.
  Interventions: Drug: cabozantinib
- Mitoxantrone/prednisone (Active Comparator): Subjects randomized to the mitoxantrone + prednisone arm will also receive placebo cabozantinib tablets.
  There will be a maximum of 10 infusions for mitoxantrone.
  Interventions: Drug: mitoxantrone; Drug: prednisone

INTERVENTIONS:
Drug: cabozantinib — Tablets taken orally once daily.
  Arms: Cabozantinib
Drug: mitoxantrone — Given by IV once every 3 weeks.
  Arms: Mitoxantrone/prednisone
Drug: prednisone — Taken twice a day orally by mouth. Commercially-obtained prednisone tablets will be over-encapsulated in order to blind identity.
  Arms: Mitoxantrone/prednisone

SUMMARY:
Bone metastases and associated pain are a major cause of morbidity and mortality in castration-resistant prostate cancer (CRPC). Most approved therapies have shown some ability to reduce soft tissue lesions but none meaningfully impacts bone metastases (as demonstrated by lack of resolution of lesions on bone scan with these agents) or the pain associated with these metastases.

This study will evaluate the effect of cabozantinib versus mitoxantrone plus prednisone on pain response and bone scan response in men with CRPC.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of castration resistant prostate cancer (serum testosterone less than 50 ng/dL).
* Evidence of bone metastasis related to prostate cancer on bone scans.
* Documented pain from bone metastases that requires opioid narcotic intervention.
* Adopted a narcotic regimen that consists of one sustained release opioid agent taken daily for chronic pain and one immediate release opioid agent for breakthrough pain.
* Received prior docetaxel and either abiraterone or MDV3100 treatment and has evidence of investigator assessed prostate cancer progression on each agent independently.
* Maintenance of LHRH agonist or antagonist unless treated with orchiectomy.
* Recovered from toxicities related to any prior treatments, unless the toxicities are clinically non significant or easily manageable.
* Adequate organ and marrow function.
* A left-ventricular ejection fraction (LVEF) of >/= 50% assessed by echocardiogram or MUGA (multigated acquisition scan).
* Capable of understanding and complying with the protocol requirements (including having the ability to access an interactive voice recognition system and self-report pain and narcotic use) and signed the informed consent form.
* Sexually active fertile patients and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 3 months after the last dose of study treatment.

Exclusion Criteria:

* Prior treatment with cabozantinib or mitoxantrone.
* Treatment with docetaxel, abiraterone, or MDV3100 in the last 2 weeks; or with any other type of cytotoxic or investigational anticancer agent in the last 2 weeks.
* Radiation therapy in the last 4 weeks (includes radiation targeting bone metastases), radionuclide treatment in the last 6 weeks, or radiation therapy to the thoracic cavity (unless radiation targets bone metastases) in the past 3 months.
* Treatment with serotonergic psychiatric medication(s) in the last 2 weeks (5 weeks for fluoxetine).
* Known brain metastases or uncontrolled epidural disease.
* Requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or FXa (coagulation factor X) inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin (above low dose levels for cardioprotection per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and prophylactic low molecular weight heparin are permitted.
* Uncontrolled, significant intercurrent illness including, but not limited to, cardiovascular disorders, gastrointestinal disorders, active infections, non-healing wounds, recent surgery.
* Clinically significant hematemesis or hemoptysis of > 0.5 teaspoon of red blood, or other signs indicative of pulmonary hemorrhage in the last 3 months, or history of other significant bleeding in the past 6 months.
* Cavitating pulmonary lesion(s) or a lesion invading or encasing a major blood vessel.
* Corrected QT interval (QTc) > 500 ms in the last 4 weeks.
* Unable to swallow capsules or tablets or tolerate infusions.
* Previously-identified allergy or hypersensitivity to components of the study treatment formulations investigator or designee.
* History of another malignancy (except non-melanoma skin cancer, adequately treated stage I colon cancer, superficial transitional carcinoma of the bladder) in the past 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2015-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (45):
  - Scottsdale, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Marina del Rey, California
  - San Diego, California
  - San Francisco, California
  - Santa Barbara, California
  - Stanford, California
  - Aurora, Colorado
  - Littleton, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Athens, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Westwood, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Buffalo, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Watertown, South Dakota
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Round Rock, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (12):
  - Concord, New South Wales
  - Darlinghurst, New South Wales
  - Kogarah, New South Wales
  - Port Macquarie, New South Wales
  - Randwick, New South Wales
  - Wahroonga, New South Wales
  - Milton, Queensland
  - South Brisbane, Queensland
  - Woolloongabba, Queensland
  - Box Hill, Victoria
  - Wodonga, Victoria
  - Subiaco, Western Australia
- Canada (4):
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
- Dublin, Ireland
- United Kingdom (12):
  - Bath, England
  - Cambridge, England
  - Leeds, England
  - London, England
  - Manchester, England
  - Metropolitan Borough of Wirral, England
  - Sutton, England
  - Aberdeen, Scotland
  - Edinburgh, Scotland
  - Glasgow, Scotland
  - Inverness, Scotland
  - Belfast

REFERENCES:
- [Derived] Thanarajasingam G, Basch E, Mead-Harvey C, Bennett AV, Mazza GL, Schwab G, Roydhouse J, Rogak LJ, Dueck AC. An Exploratory Analysis of the "Was It Worth It?" Questionnaire as a Novel Metric to Capture Patient Perceptions of Cancer Treatment. Value Health. 2022 Jul;25(7):1081-1086. doi: 10.1016/j.jval.2021.11.1368. Epub 2022 Jan 3. PMID 35779938
- [Derived] Mazza GL, Petersen MM, Ginos B, Langlais BT, Heon N, Gounder MM, Mahoney MR, Zoroufy AJ, Schwartz GK, Rogak LJ, Thanarajasingam G, Basch E, Dueck AC. Missing data strategies for the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) in Alliance A091105 and COMET-2. Qual Life Res. 2022 Apr;31(4):1069-1080. doi: 10.1007/s11136-021-02968-1. Epub 2021 Aug 21. PMID 34420143
- [Derived] Basch E, Becker C, Rogak LJ, Schrag D, Reeve BB, Spears P, Smith ML, Gounder MM, Mahoney MR, Schwartz GK, Bennett AV, Mendoza TR, Cleeland CS, Sloan JA, Bruner DW, Schwab G, Atkinson TM, Thanarajasingam G, Bertagnolli MM, Dueck AC. Composite grading algorithm for the National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Clin Trials. 2021 Feb;18(1):104-114. doi: 10.1177/1740774520975120. Epub 2020 Dec 1. PMID 33258687
- [Derived] Dueck AC, Scher HI, Bennett AV, Mazza GL, Thanarajasingam G, Schwab G, Weitzman AL, Rogak LJ, Basch E. Assessment of Adverse Events From the Patient Perspective in a Phase 3 Metastatic Castration-Resistant Prostate Cancer Clinical Trial. JAMA Oncol. 2020 Feb 1;6(2):e193332. doi: 10.1001/jamaoncol.2019.3332. Epub 2020 Feb 13. PMID 31556911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 15 March 2012, Data cut off date: 06 October 2014. The study was terminated by the Sponsor after 119 subjects were enrolled which was less than the planned sample size of 246 subjects.
Groups:
- Cabozantinib: Subjects randomized to the cabozantinib arm will also receive placebo mitoxantrone injections (color-matched with methylene blue) and placebo prednisone capsules.
  Cabozantinib (XL184) 60 mg tablets taken orally once daily and mitoxantrone-matched placebo infusion every 3 weeks (maximum of 10 infusions) plus prednisone-matched placebo capsules orally twice daily.
- Mitoxantrone/Prednisone: Subjects randomized to the mitoxantrone + prednisone arm will also receive placebo cabozantinib tablets.
  Mitoxantrone (12mg/m^2) given by IV once every 3 weeks (maximum of 10 infusions) plus prednisone-matched placebo capsules orally twice daily.
Period: Overall Study
Arm/Group | Cabozantinib | Mitoxantrone/Prednisone
Started (Randomized) | 61 | 58
Completed (Subjects still on study treatment at data cut-off date) | 8 | 3
Not Completed | 53 | 55
Not completed — No longer receiving clinical benefit | 36 | 28
Not completed — Adverse Event | 10 | 15
Not completed — Withdrawal by Subject | 5 | 8
Not completed — No study treatment given | 1 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib | Mitoxantrone/Prednisone | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Customized [Number; unit: participants]
  <65 years | 24 | 26 | 50
  65 to <75 years | 30 | 26 | 56
  75 to <85 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 58 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 57 | 57 | 114
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Black/African-American | 8 | 3 | 11
  Multiple | 1 | 0 | 1
  White | 49 | 51 | 100
  Not Reported | 0 | 1 | 1
  Other | 1 | 0 | 1
Geographic Region [Number; unit: participants]
  North America | 44 | 36 | 80
  Europe | 8 | 13 | 21
  Asia | 9 | 9 | 18
ECOG Performance Status (per IVRS/IWRS) [Number; unit: participants]
  0-1 (normal to symptoms, but ambulatory) | 53 | 52 | 105
  ≥2 (ambulatory to incapable of self-care/death) | 8 | 6 | 14
Randomization Stratification Factors (per IVRS/IWRS) [Number; unit: participants]
  ECOG = 0-1 and prior cabazitaxel: yes | 18 | 18 | 36
  ECOG = 0-1 and prior cabazitaxel: no | 35 | 34 | 69
  ECOG ≥ 2 and prior cabazitaxel: yes | 7 | 6 | 13
  ECOG ≥ 2 and prior cabazitaxel: no | 1 | 0 | 1
Time from initial diagnosis to randomization [Median (Full Range); unit: years] | 4.7 [0 to 18] | 5.3 [0 to 16] | 5.0 [0 to 18]
Gleason score at diagnosis (Primary + Secondary) [Number; unit: participants] — The Gleason score is used to define prostate cancer prognosis by histologic grading with scores ranging from 2 to 10. A higher Gleason score indicates a more aggressive form of prostate cancer with a worse prognosis.
  participants
    <7 | 2 | 4 | 6
    7 | 17 | 21 | 38
    >7 | 40 | 28 | 68
    Unknown | 2 | 4 | 6
    Missing | 0 | 1 | 1
Prior prostate surgery/procedure [Number; unit: participants] — Baseline radical prostatectomy with and without retropubic with pelvic lymphadenectomy measures are provided.
  participants
    Transurethral resection of the prostate (TURP) | 8 | 6 | 14
    Radical prostatectomy - with | 17 | 13 | 30
    Radical prostatectomy - without | 3 | 2 | 5
    Cyrosurgery | 0 | 1 | 1
    Bilateral orchiectomy | 4 | 2 | 6
    Other | 55 | 52 | 107
Bone-scan lesion area (BSLA) [Median (Full Range); unit: mm^2] | 72865.0 [0 to 251469] | 72702.5 [679 to 281936] | 72865.0 [0 to 281936]
Sites of prostate cancer metastasis [Number; unit: participants]
  Bone | 61 | 58 | 119
  Lymph node | 29 | 18 | 47
  Visceral (soft tissue; liver) | 8 | 8 | 16
  Visceral (soft tissue; lung) | 2 | 5 | 7
  Other soft tissue | 7 | 3 | 10
Pain score (BPI Item 3) during Run-In Stage [Median (Full Range); unit: units on a scale] — During the Run-In State, subjects will self-report pain by phone via an interactive voice response system (IVRS) daily for 7 days and record analgesic medication information on a paper pain medication diary. Each day of the reporting periods, subjects will report their worst pain intensity and their average pain intensity over a 24-hour period using an 11-point numerical rating system (NRS) (ranging from 0 to 10, with 0 representing "No Pain," and 10 representing "Pain as Bad as You Can Imagine").
  units on a scale | 6.00 [4.0 to 8.0] | 6.14 [4.0 to 8.0] | 6.00 [4.0 to 8.0]
Pain score (BPI Item 3) during Run-In Stage [Number; unit: participants] — During the Run-In State, subjects will self-report pain by phone via an interactive voice response system (IVRS) daily for 7 days and record analgesic medication information on a paper pain medication diary. Each day of the reporting periods, subjects will report their worst pain intensity and their average pain intensity over a 24-hour period using an 11-point numerical rating system (NRS) (ranging from 0 to 10, with 0 representing "No Pain," and 10 representing "Pain as Bad as You Can Imagine").
  participants
    4-5 | 10 | 15 | 25
    >5-6 | 22 | 13 | 35
    >6-7 | 18 | 15 | 33
    >7-8 | 11 | 15 | 26
Number of prior anticancer agents [Count of Participants; unit: Participants]
  2 | 0 | 3 | 3
  3 | 6 | 4 | 10
  4 | 20 | 14 | 34
  ≥5 | 35 | 37 | 72
Prior cabazitaxel (per IVRS/IWRS) [Count of Participants; unit: Participants]
  Yes | 25 | 24 | 49
  No | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Pain Response at Week 6 Confirmed at Week 12, Week 12 Reported
Description: The pre-specified primary analysis of Pain Response at Week 6 confirmed at Week 12 was defined as ≥ 30% from baseline in the average daily worst pain intensity score during a 7-day reporting period, with neither a concomitant increase in average daily use of any opioid narcotic type, nor addition of any new opioid narcotic type, relative to baseline. Pain Progression at a given time point is defined as ≥ 30% increase compared with baseline in the average daily worst pain intensity score during a 7-day reporting period or either an increase in the average daily use of any type of opioid narcotic or addition of a new opioid narcotic type compared with baseline.
Time Frame: Pain response was measured at Week 6 and Week 12 by self-reports of subjects
Population: The primary analysis of pain response was based on the Intent to Treat (ITT) population of 119 participants (61 cabozantinib, 58 mitoxantrone plus prednisone).
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Cabozantinib | Mitoxantrone/Prednisone
Number analyzed (Participants) | 61 | 58
percentage of responders | 15 [5.9 to 24] | 17 [7.5 to 27]
Statistical Analysis 1: Comparison: Cabozantinib vs Mitoxantrone/Prednisone; Test type: Superiority or Other; p = 0.773, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel (CMH) was stratified by the Eastern Cooperative Oncology Group performance status and prior cabazitaxel use

2. Secondary Outcome: Bone Scan Response (BSR)
Description: BSR is defined as >=30% in the bone scan lesion area (BSLA) compared with baseline. Bones scans were evaluated by an independent radiology facility (IRF) for response.
Time Frame: BSR was measured at the end of Week 12 as determined by the IRF
Population: Analysis was conducted on the randomized ITT population (61 cabozantinib, 58 mitoxantrone plus prednisone) for BSR at Week 12.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Cabozantinib | Mitoxantrone/Prednisone
Number analyzed (Participants) | 61 | 58
percentage of responders | 31 [20 to 43] | 5.2 [0 to 11]
Statistical Analysis 1: Comparison: Cabozantinib vs Mitoxantrone/Prednisone; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel (CMH) Test was stratified by baslined Eastern Cooperative Oncology Group performance status and prior cabazitaxel use

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death (due to any cause). Participants that had not died were censored at last known date alive. The analyses for OS occurred after 78/196 deaths (40% of the total required for the pre-specified primary analysis of OS). The data cut-off date was 06 October 2014. Median OS was calculated using Kaplan-Meier estimates.
Time Frame: OS was measured at the time of randomization until 78 deaths
Population: The Intent to Treat (ITT) population was used and included 119 randomized subjects (61 cabozantinib, 58 mitoxantrone plus prednisone) at the time of primary analysis (data cut off date: 06 October 2014).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib | Mitoxantrone/Prednisone
Number analyzed (Participants) | 61 | 58
months | 9.0 [6.80 to 11.56] | 7.9 [5.26 to 9.10]
Statistical Analysis 1: Comparison: Cabozantinib vs Mitoxantrone/Prednisone; Test type: Superiority or Other; p = 0.121, Log Rank; The Log-Rank Test was stratified by baseline Eastern Cooperative Oncology Group performance status and prior cabazitaxel use; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.44 to 1.10]

ADVERSE EVENTS:
Time Frame: Up to 95 weeks
Description: The safety data includes subjects who were randomized and treated with at least one dose of the study treatment. Of 119 patients, 61 were randomized to receive cabozantinib and 58 mitoxantrone plus prednisone. The Safety population included 117 subjects (60 cabozantinib, 57 mitoxantrone plus prednisone).
Arm/Group | Cabozantinib | Mitoxantrone/Prednisone
Serious Adverse Events (participants affected / at risk) | 16/60 | 15/57
Other Adverse Events (participants affected / at risk) | 60/60 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=60) | Mitoxantrone/Prednisone (N=57)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=60) | Mitoxantrone/Prednisone (N=57)
Nausea (Gastrointestinal disorders) | 38 | 24
Fatigue (General disorders) | 34 | 27
Decreased appetite (Metabolism and nutrition disorders) | 28 | 23
Diarrhoea (Gastrointestinal disorders) | 27 | 17
Weight decreased (Investigations) | 25 | 8
Constipation (Gastrointestinal disorders) | 24 | 19
Vomiting (Gastrointestinal disorders) | 23 | 19
Hypertension (Vascular disorders) | 18 | 0
Asthenia (General disorders) | 14 | 4
Depression (Psychiatric disorders) | 14 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 4
Aspartate aminotransferase increased (Investigations) | 12 | 2
Alanine aminotransferase increased (Investigations) | 10 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 9 | 4
Insomnia (Psychiatric disorders) | 9 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 | 0
Blood alkaline phosphatase increased (Investigations) | 8 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Oral pain (Gastrointestinal disorders) | 7 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 2
Hypothyroidism (Endocrine disorders) | 6 | 1
Neutrophil count decreased (Investigations) | 6 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 0
Glossodynia (Gastrointestinal disorders) | 4 | 0
Lymphocyte count decreased (Investigations) | 4 | 0
Proteinuria (Renal and urinary disorders) | 4 | 0
Blister (Skin and subcutaneous tissue disorders) | 3 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Depressed mood (Psychiatric disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Musculoskeletal stiffness (Metabolism and nutrition disorders) | 3 | 0
Pallor (Vascular disorders) | 3 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 0
Retching (Gastrointestinal disorders) | 3 | 0
Sinusitis (General disorders) | 3 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Enrollment was stopped before planned study population size of 246 was reached (only 119 enrolled).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements with investigators vary; constant is our right to review results communications prior to public release, and embargo communications for a period of ≤60 days from submittal for review. We do not prohibit investigators from publishing, but we may require previously undisclosed confidential information, other than study results, to be removed from publications, and single-center publications are postponed until after publication of the trial's primary multicenter publication.